CLINICAL TRIAL: NCT05492292
Title: Long-term Effects of SARS-CoV-2 on the Central Nervous System and One-year Follow-up of "Long COVID-19" Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Bernard Dachy, Head of Neurology Department, Brugmann University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUB-Neuro-Covid Long
Record Dates: First submitted 2022-08-02; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Long Covid19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Long Covid19 patient group (Experimental): Patients with Long Covid19 undergoing perfusion brain scintigraphy
  Interventions: Diagnostic Test: Perfusion brain scintigraphy imaging

INTERVENTIONS:
Diagnostic Test: Perfusion brain scintigraphy imaging — The cerebral perfusion scintigraphy via a SPECT examination aims to analyze the cerebral blood flow and detect possible lesions or inflammations.

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is the seventh coronavirus known to infect humans, and causing coronavirus disease 2019 (COVID-19). . Since its emergence in December 2019, in Wuhan, China, SARS-CoV-2 has led to a global pandemic with almost 188 million cases and 4 million COVID-19 related deaths reported. Although initially considered as a predominantly acute respiratory illness, it soon became apparent that COVID-19 could also produce neurological manifestations and severe neurological complications. During the acute phase of SARS-CoV-2 infection, about 36% of cases develop neurological symptoms of which 25% can be attributed to the direct involvement of the central nervous system.

There are increasing reports of central and peripheral nervous system involvement. Acute neurological manifestations reported, include, but are not limited to: anosmia, dysgeusia, stroke, encephalomyelitis, meningo-encephalitis, posterior reversible encephalopathy, acute necrotizing encephalopathy, new onset seizures and Guillain-Barre syndrome.

However, one of the most perplexing aspects of SARS-CoV-2 is that two to four months after their initial (mostly apparently mild) infection, some COVID-19 patients still present a constellation of more chronic neurological symptoms colloquially known as "long COVID-19" syndrome. In these patients, COVID-19 appears to affect long-term brain function and patients have functional complaints as dyspnea, hyposmia/anosmia, dysgeusia/ageusia, but also, and more importantly, memory and cognitive impairment, pain, deadening fatigue, and alterations in sleeping-pattern/insomnia, all of them correlated with typical 18F-FDG brain PET scan abnormalities.

At the beginning of the pandemic, the medical world was not expecting the phenomenon of COVID-19 patients developing persistent neurologically symptoms. However, more than one year after the pandemic, multiple waves of the "long COVID-19" syndrome may be expected to occur worldwide. To face the long tail impact of the COVID-19 pandemic on public health and its social and economic consequences on our society, future research urgently needs to be dedicated to these "long COVID-19" patients in an attempt to determine, understand and manage their symptoms.

A lot of "long COVID-19" patients are desperately searching for help. This project found his origin in the fact that suddenly many patients spontaneously presented with a similar constellation of persistent (chronic) symptoms, months after they had (mostly mild) COVID-19, with many of them being relatively young, without underlying health problems, but unable to work due to cognitive impairment. During the entire study, the opinion and feelings of these patients will be taken in account, all the more so because the majority of these patients were initially left behind.

The primary objective of this study is to determine the different types of neurological dysfunction and clinical manifestations of the "long COVID-19" syndrome and to correlate them to abnormalities/signs on cerebral perfusion scintigraphy. Furthermore, the investigators aim to determine and validate a specific imaging biomarker of post-COVID-19 encephalopathy.

The secondary objective of this study is to determine the best therapeutic modality to treat and improve prognosis of patients with "long COVID-19" syndrome with defined central nervous system impairment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Physically and mentally able to fill out questionnaires;
* Suspicion and/or confirmation of COVID-19 infection, managed on an out- or inpatient (COVID-19 ward or ICU) basis;
* Residual symptoms at 8 weeks or more after initial SARS-CoV-2 infection.

Exclusion Criteria:

* Diagnosed with a neurological syndrome e.g. Parkinson disease, Alzheimer disease, … before SARS-CoV-2 infection;
* Known Dementia or mild cognitive impairment before SARS-CoV-2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference (1 year versus baseline) in the distribution of hypo-perfused areas in the brain as assessed by cerebral perfusion scintigraphy. | 1 year
  SPECT data were acquired using a standardized protocol. For focal abnormalities of increased or decreased uptake, the anatomical location was described.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Dominique Gazagnes, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium